CLINICAL TRIAL: NCT01983085
Title: ProNOx 2 - A Clinical Study of Superficial Partial Thickness Wound Treatment With an Oxides of Nitrogen Generating Gel Dressing
Brief Title: Nitric Oxide Generating Gel Dressing in Patients With Superficial Partial Thickness Wounds
Acronym: ProNOx2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was paused initially pending a review of the study design. The decision was then taken not to resume the study.
Sponsor: Edixomed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDX 120
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Superficial Partial Thickness Burn; Skin Graft; Complications
Keywords: Nitric Oxide Dressing; Nitric oxide; Superficial partial thickness wound; Burns; Skin graft donor sites; Improved healing; Vasodilation; Angiogenesis; Anti-microbial
MeSH Terms: conditions — Burns; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPT Burn Wound (Other): Each wound will be divided into 2 with half the wound being treated with the NOx dressing and the other half with standard of care
  Interventions: Device: NOx dressing; Device: Standard of Care
- SPT graft donor site (Other): Each wound will be divided into 2 with half the wound being treated with the NOx dressing and the other half with standard of care
  Interventions: Device: NOx dressing; Device: Standard of Care

INTERVENTIONS:
Device: NOx dressing — The NOx dressing should be changed at least every 2 days.
Device: Standard of Care — Dressing changed as per normal clinical practice

SUMMARY:
This is a study to assess the safety and efficacy of a nitric oxide (NOx) generating dressing on superficial partial thickness (SPT) wounds. Nitric oxide has a range of effects on the body including vasodilation and angiogenesis. It is also a potent antimicrobial. This 160 patient, randomised, controlled clinical study will assess the ability of a simple 2 part, NOx generating dressing to improve healing in SPT burn wounds and SPT skin graft donor site wounds compared to standard of care.

DETAILED DESCRIPTION:
This is a clinical study of a new wound dressing for superficial partial thickness (SPT) wounds. The dressing consists of 2 stable layers that when placed together release Nitric Oxide. In preclinical studies NOx delivery has caused significant vasodilation, angiogenesis and demonstrated potent anti-microbial activity.

This is a multi-centre, 160 patient, randomised, controlled study. There are 2 arms to the study. 80 patients will have treatment applied to a SPT burn wound and 80 patients will have treatment applied to a SPT graft donor site wound.

The controls will be intra-individual. Each patient will have their wound divided into 2, half of the wound being treated with the NOx dressing, the other half treated with standard of care. The positioning of the dressings will be randomised.

The NOx dressing will be changed at least every 2 days and the standard of care changed according to normal clinical practice and patients will be treated until the wound is healed.

The study will evaluate:

* The size of the wound
* Eepithelialisation
* Trans-epidermal water loss
* Infection status.

There will be 3 and 12 month follow up with assessment of scarring.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a Superficial Partial Thickness wound (2a) either from a thermal injury or from a skin graft donor site under the care of St. Andrews service, within the recruitment timeline.
* Wound area to be treated in study must be less than 5% of total body surface area (TBSA).
* Patients aged over 12 months and up to and including 80 years old.
* Informed Consent

Exclusion Criteria:

* Any inclusion criteria not met
* Unwilling to consent to investigation/ unable to provide consent
* Wounds deeper than superficial partial thickness (2b, 3 and 4)
* Chemical /Electrical burns
* Already having received silver sulfadiazine
* Disease that could affect wound healing
* Previous participation in the study
* Females who are pregnant or breast-feeding.
* Relative, spouse or employee of the investigational site
* Known multiple allergic disorders
* Skin disorders
* Facial burns
* Patients who have taken part in any investigational studies within the last 30 days prior to participation.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Average number of days until healing (defined as 95% epithelisation) in SPT wounds treated with conventional Mepitel® dressing vs. investigational nitric oxide generating gel dressing | From randomisation and first application of the dressing, patients are assessed every 2 days until 95% epithelialisation occurs

SECONDARY OUTCOMES:
Assessment of healing by blinded evaluation of photographs | Every 2 days from baseline until 95% epithelialisation occurs
Cosmetic Outcomes measured using both the Vancouver Scar Scale and the Patient Observer Scar Assessment Scale | 3 and 12 months post healing
Colonisation of wounds | Baseline and every 2 days therafter until 95% epithelialisation occurs
  Wound swabs will be taken at every patient visit, every 2 days, until 95% epithelialisation occurs.
Tolerance and safety of the dressing | Baseline and every 2 days thereafter
  Assessment of reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stewart, PhD, Principal Investigator — Queen Mary University London
Locations (2):
- United Kingdom (2):
  - St Andrew's Centre for Plastic Surgery and Burns, Broomfield Hospital, Chelmsford, Essex
  - Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow Royal Infirmary,, Glasgow